CLINICAL TRIAL: NCT05736757
Title: Application of tPA in Suprachoroidal and Subretinal Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0178
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-07

CONDITIONS: Ocular Trauma
Keywords: suprachoroidal hemorrhage; subretinal hemorrhage
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Randomly divided into control group (without tissue fibrinogen activator) or drug group (injection of 50 ug tissue fibrinogen activator into the suprachoroidal cavity or subretinal space ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group (no tissue fibrinogen activator)
- Drug group (Experimental): Drug group (injection of 50 ug tissue fibrinogen activator into the suprachoroidal cavity or subretinal space )
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — Injection of 50 ug tissue plasminogen activator into the suprachoroidal cavity or subretinal space to assist in bleeding liquefaction
  Arms: Drug group

SUMMARY:
Severe ocular rupture may be accompanied by suprachoroidal hemorrhage, or subretinal hemorrhage, or with suprachoroidal hemorrhage and subretinal hemorrhage. The suprachoroidal hemorrhage needs to be drained as soon as possible. In the process of waiting for the spontaneous liquefaction of hemorrhage, uncontrollable elevated intraocular pressure may occur, resulting in optic nerve injury, optic nerve atrophy, and visual loss. Tissue plasminogen activator can promote the liquefaction of blood clots. Studies have found that local application of tissue plasminogen activator in the suprachoroidal space can promote the liquefaction of the hemorrhage. Local application of tissue fibrinogen activator under the retina can promote the liquefaction of subretinal hemorrhage.

DETAILED DESCRIPTION:
Severe ocular rupture may be accompanied by suprachoroidal hemorrhage, or subretinal hemorrhage, or with suprachoroidal hemorrhage and subretinal hemorrhage. The suprachoroidal hemorrhage needs to be drained as soon as possible. The traditional treatment method needs to wait for the spontaneous liquefaction of the suprachoroidal hemorrhage, and then perform scleral incision to drain the liquefied suprachoroidal hemorrhage. However, in the process of waiting for the spontaneous liquefaction of suprachoroidal hemorrhage, uncontrollable elevated intraocular pressure may occur, resulting in optic nerve injury, optic nerve atrophy, and visual loss. In addition, if the suprachoroidal hemorrhage is not completely liquefied, it will not be completely drained, which will lead to choroidal function damage, low intraocular pressure and eyeball atrophy.

Severe ocular rupture can be accompanied by a large amount of subretinal hemorrhage. The traditional treatment is to open the retina in a large area and drain the subretinal hemorrhage. However, extensive retinal incision has great damage, vitreoretinal proliferation often occurs after surgery, leading to recurrent retinal detachment, large area of choroid exposure, low intraocular pressure, and atrophy of the eye.

Tissue plasminogen activator can promote the liquefaction of blood clots. Studies have found that local application of tissue plasminogen activator in the suprachoroidal space can promote the liquefaction of the hemorrhage near the suprachoroidal space, and can drain the hemorrhage of the suprachoroidal space smoothly and completely in the early stage. Local application of tissue plasminogen activator under the retina can promote the liquefaction of subretinal hemorrhage. Through small retinal incision, subretinal hemorrhage can be completely drained, the scope of retinal incision can be reduced, vitreoretinal proliferation can be reduced, and the occurrence of recurrent retinal detachment after surgery can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe ocular rupture accompanied by suprachoroidal hemorrhage, or subretinal hemorrhage, or with suprachoroidal hemorrhage and subretinal hemorrhage

Exclusion Criteria:

* Rupture of eyeball accompanied by a small amount of suprachoroidal hemorrhage or a small amount of subretinal hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | through study completion, an average of 2 year
  Best corrected visual acuity

SECONDARY OUTCOMES:
Intraocular pressure | through study completion, an average of 2 year
  Intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- See also: Tissue plasminogen activator-assisted vitrectomy for ruptured eye with suprachoroidal hemorrhage — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=22949914&query_hl=1
- See also: Tissue plasminogen activator-assisted vitrectomy in the early treatment of acute massive suprachoroidal hemorrhage complicating cataract surgery — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=29376008&query_hl=1
- See also: Recombinant tissue plasminogen activator in the treatment of suprachoroidal hemorrhage — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=21383941&query_hl=1
- See also: Tissue plasminogen activator in the treatment of vitreoretinal diseases — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=10749314&query_hl=1
- See also: Treatment of suprachoroidal hemorrhage with tissue plasminogen activator — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=9486552&query_hl=1
- See also: Treatment of experimental suprachoroidal hemorrhage with intravenous tissue plasminogen activator — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=2115030&query_hl=1